CLINICAL TRIAL: NCT03250286
Title: Role of EUS in High Risk of Choledocholithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woo Hyun Paik (Other)
Responsible Party: Sponsor-Investigator, Woo Hyun Paik, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1705-070-854
Record Dates: First submitted 2017-07-18; First posted 2017-08-15 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-ERCP group (Experimental): EUS is performed first, and when the examiner finds bile duct stone in the EUS examination, ERCP is performed to remove the stone.
  Interventions: Device: EUS; Device: ERCP
- ERCP group (Active Comparator): ERCP without EUS is performed in all patients.
  Interventions: Device: ERCP

INTERVENTIONS:
Device: EUS — Endoscopic ultrasound (EUS) is performed with radial scanning echo endoscope (Olympus GF UE260) by four endosonographers.
  EUS examination is performed first, and if there is choledocholith, ERCP is performed.
  Arms: EUS-ERCP group
Device: ERCP — Endoscopic retrograde cholangiopancreatography (ERCP) is performed with duodenoscope (Olympus JF-260V or TJF-260V) by four endoscopists.
  * In the EUS-ERCP group, ERCP is used to remove bile duct stones diagnosed via EUS. Therefore, only ERCP is performed in patients with choledocholithiasis in EUS.
  * In the ERCP group, diagnosis and treatment of bile duct stones are performed with ERCP.

SUMMARY:
The aim of this study is to demonstrate that patients with high risk of choledocholithiasis who undergo ERCP only for patients with choledocholith in the EUS examination[EUS-ERCP group] have less negative outcomes (including false-negative results and procedure-related complications) than patients who undergo ERCP in all patients with high risk of choledocholithiasis[ERCP group]. The primary outcome is the incidence of negative outcomes (including false-negative results and procedure-related complications) in both groups. The secondary outcomes included days of hospitalization and the rate of diagnostic ERC.

DETAILED DESCRIPTION:
Several studies have shown that EUS testing prior to ERCP may reduce ERCP complications in patients with intermediate-risk choledocholithiasis. In other words, this results obtained by not performing ERCP in patients without choledocholith in the EUS examination. However, to the best of our knowledge, no prospective study has been conducted on the role of EUS in patients with high risk of choledocholithiasis. Therefore, we investigate the role of EUS screening in patients with high risk of choledocholithiasis. We compare the negative outcomes (including false negative and procedure-related complications of EUS and ERCP) of the 'EUS-ERCP group' in which ERCP is performed when necessary after the EUS examination and the 'ERCP group' in which ERCP is performed in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal CT or US showed a common bile duct diameter > 6mm (>8mm in patients with previous cholecystectomy) and elevated total bilirubin from 1.8mg/dL to less than 4.0mg/dL

Exclusion Criteria:

* Severe mental illness
* Severe co-morbidity (ESRD, Advanced COPD, severe Heart failure, poorly controlled blood sugar)
* Pregnancy
* Pancreatic cancer or suspected malignant tumor of the biliary tract
* Acute pancreatitis
* Patient who has confirmed biliary stones in abdominal ultrasonography or CT
* Severe cholangitis according to TG 18 guideline
* Total bilirubin > 4mg/dL
* Patients who have difficulty with EUS or ERCP due to previous gastric surgery (Billroth II or TG with R-en-Y)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Any negative outcomes related to either a false-negative diagnosis of choledocholithiasis or the endoscopic procedure | 6 months after randomization
  Negative outcomes associated with a false-negative diagnosis of choledocholithiasis were defined as follows: 1) diagnosis of choledocholithiasis during follow-up or 2) hospitalization for a condition likely associated with choledocholithiasis, such as biliary pancreatitis, cholangitis, or obstructive jaundice. Negative outcomes of endoscopic procedures were assessed according to the ASGE lexicon

SECONDARY OUTCOMES:
Length of hospital stay | 6 months after randomization
  Length of hospital stay

OTHER OUTCOMES:
The rate of diagnostic ERC (Endoscopic retrograde cholangiography) | 6 months after randomization
  The diagnostic ERC was defined as any ERC procedures in which no stone or sludge was removed during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Hyun Paik, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Maple JT, Ben-Menachem T, Anderson MA, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Strohmeyer L, Dominitz JA. The role of endoscopy in the evaluation of suspected choledocholithiasis. Gastrointest Endosc. 2010 Jan;71(1):1-9. doi: 10.1016/j.gie.2009.09.041. No abstract available. PMID 20105473
- [Background] He H, Tan C, Wu J, Dai N, Hu W, Zhang Y, Laine L, Scheiman J, Kim JJ. Accuracy of ASGE high-risk criteria in evaluation of patients with suspected common bile duct stones. Gastrointest Endosc. 2017 Sep;86(3):525-532. doi: 10.1016/j.gie.2017.01.039. Epub 2017 Feb 4. PMID 28174126
- [Background] Tse F, Liu L, Barkun AN, Armstrong D, Moayyedi P. EUS: a meta-analysis of test performance in suspected choledocholithiasis. Gastrointest Endosc. 2008 Feb;67(2):235-44. doi: 10.1016/j.gie.2007.09.047. PMID 18226685
- [Background] Garrow D, Miller S, Sinha D, Conway J, Hoffman BJ, Hawes RH, Romagnuolo J. Endoscopic ultrasound: a meta-analysis of test performance in suspected biliary obstruction. Clin Gastroenterol Hepatol. 2007 May;5(5):616-23. doi: 10.1016/j.cgh.2007.02.027. PMID 17478348
- [Background] De Castro VL, Moura EG, Chaves DM, Bernardo WM, Matuguma SE, Artifon EL. Endoscopic ultrasound versus magnetic resonance cholangiopancreatography in suspected choledocholithiasis: A systematic review. Endosc Ultrasound. 2016 Mar-Apr;5(2):118-28. doi: 10.4103/2303-9027.180476. PMID 27080611
- [Background] Polkowski M, Regula J, Tilszer A, Butruk E. Endoscopic ultrasound versus endoscopic retrograde cholangiography for patients with intermediate probability of bile duct stones: a randomized trial comparing two management strategies. Endoscopy. 2007 Apr;39(4):296-303. doi: 10.1055/s-2007-966264. PMID 17427065
- [Background] Adams MA, Hosmer AE, Wamsteker EJ, Anderson MA, Elta GH, Kubiliun NM, Kwon RS, Piraka CR, Scheiman JM, Waljee AK, Hussain HK, Elmunzer BJ. Predicting the likelihood of a persistent bile duct stone in patients with suspected choledocholithiasis: accuracy of existing guidelines and the impact of laboratory trends. Gastrointest Endosc. 2015 Jul;82(1):88-93. doi: 10.1016/j.gie.2014.12.023. Epub 2015 Mar 16. PMID 25792387